CLINICAL TRIAL: NCT01160640
Title: The Importance of Anti-anaerobic Therapy for Acute PID
Brief Title: The Importance of Anti-anaerobic Therapy for Acute Pelvic Inflammatory Disease (PID)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harold Wiesenfeld (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Harold Wiesenfeld, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO10010112; 1U19AI084024-01 (NIH)
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Pelvic Inflammatory Disease
Keywords: PID; Pelvic Inflammatory Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — Ceftriaxone; Doxycycline; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceftriaxone/Doxycycline/Placebo Oral Cap (Placebo Comparator): ceftrixone 250mg IM single dose plus doxycycline 100 mg PO bid x 14 days plus placebo oral capsule PO bid x 14 days
  Interventions: Drug: Ceftriaxone; Drug: Doxycycline; Drug: Placebo Oral Capsule
- Ceftriaxone, Doxycycline, Metronidazole (Active Comparator): ceftriaxone 250 mg IM single dose plus doxycycline 100 mg PO bid x 14 days plus metronidazole 500 mg PO bid x 14 days
  Interventions: Drug: Ceftriaxone; Drug: Doxycycline; Drug: Metronidazole

INTERVENTIONS:
Drug: Ceftriaxone — ceftrixone 250mg IM single dose
  Other Names: Rocephin
Drug: Doxycycline — Doxycycline 100 mg PO bid x 14 days
Drug: Metronidazole — metronidazole 500 mg PO bid x 14 days
  Other Names: Flagyl
  Arms: Ceftriaxone, Doxycycline, Metronidazole
Drug: Placebo Oral Capsule — placebo oral capsule PO bid x 14 days
  Arms: Ceftriaxone/Doxycycline/Placebo Oral Cap

SUMMARY:
This study is a randomized placebo-controlled trial comparing two antibiotic treatment regimens for acute PID. Women with acute PID will be randomized to one of two treatment regimens: 1) a single intramuscular dose of ceftriaxone 250 mg, doxycycline 100 mg orally twice a day for 14 days, along with placebo tablets orally twice a day for 14 days or 2) same doses of ceftriaxone and doxycycline, and metronidazole 500 mg orally twice a day for 14 days. The primary objective is to compare the eradication of anaerobic organisms from the upper genital tract between women who receive standard outpatient antibiotic treatment to those who receive standard outpatient treatment along with a two-week course of metronidazole.

DETAILED DESCRIPTION:
This study is a randomized placebo-controlled trial comparing two antibiotic treatment regimens for acute PID. Women with acute PID will be randomized to one of two treatment regimens. One group of women will receive a single intramuscular dose of ceftriaxone 250 mg, doxycycline 100 mg orally twice a day for 14 days, along with placebo tablets orally twice a day for 14 days. The second group of women will receive the same doses of ceftriaxone and doxycycline, and metronidazole 500 mg orally twice a day for 14 days. The primary objective is to compare the eradication of anaerobic organisms from the upper genital tract in women with acute PID who receive standard outpatient antibiotic treatment to the eradication of these organisms from the upper genital tract in women who receive standard outpatient treatment along with a two-week course of metronidazole. Women will be followed for one month for clinical outcomes, and will undergo assessment for clearance of microorganisms from the upper genital tract. Our hypothesis is that an antibiotic treatment regimen that includes anaerobic coverage will more effectively clear anaerobic organisms from the endometrium in women with acute PID compared to a standard antibiotic treatment regimen lacking effective antibiotic coverage against anaerobes.

ELIGIBILITY:
Inclusion Criteria:

Women must meet all of the following inclusion criteria:

1. Age 15-40 at the time of enrollment (Note: Participants between the ages of 15-17 will require written informed consent from parent/legal guardian. Written assent will also be obtained from the minor)
2. Acute PID, defined by symptoms and signs guided by current CDC guidelines:50

   1. Current symptoms of lower abdominal or pelvic pain (present for ≤30 days) AND
   2. Cervical motion tenderness AND/OR uterine tenderness AND/OR adnexal tenderness on pelvic examination
3. Ability to provide written informed consent

Exclusion Criteria:

Women with any of the following will be ineligible to participate:

1. Pregnant or nursing a baby (Note: a urine pregnancy test will be done at enrollment. Result must be negative to participate in the study.)
2. Uterine procedure (e.g. dilation and curettage, abortion) or miscarriage within the past 6 weeks.
3. Allergy to any of the study medications (cephalosporins, doxycycline, or metronidazole) or Type 1 hypersensitivity allergic reaction to penicillin for those with unknown tolerance to cephalosporins.
4. Systemic or vaginal antibiotic therapy in the preceding 7 days
5. Requires inpatient PID therapy (per the current CDC guidelines)50
6. Inability to obtain an endometrial biopsy at enrollment
7. Known inability to comply with the follow-up visits
8. Prior hysterectomy
9. Menopause (including natural menopause defined as lack of menses for 12 consecutive months [in the absence of pregnancy] and surgical menopause defined as a woman who has had both ovaries removed)
10. Inability to swallow pills
11. Not willing to refrain from alcohol during the two week treatment period (and two additional days following completion of study medication)
12. Other condition present at enrollment that requires additional antibiotic treatment
13. Current use of any of the following medications:

    * Anticoagulants, coumarin- or indandione-derivative: warfarin
    * cimetidine (Tagamet)
    * Disulfiram
    * Seizure medications including: phenytoin (Dilantin), carbamezapine (Tegretol), barbiturates (i.e. Phenobarbital)
    * Lithium
    * Immunosuppressive drugs including: cyclosporine, amprenavir
    * Antacids, minerals or bismuth subsalicylate (Pepto Bismol)
14. Any condition, in the opinion of the investigator that would interfere with the participant's safety or with study outcomes
15. Participation in any study involving an investigational product in the past 30 days or anticipation of participation in any study using an investigational product in the next 30 days
16. Previous participation in this study
17. Evidence of a tuboovarian abscess

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 233 (Actual)
Dates: Start 2010-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold C Wiesenfeld, MD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Allegheny County Health Department Sexually Transmitted Diseases Clinic, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiesenfeld HC, Meyn LA, Darville T, Macio IS, Hillier SL. A Randomized Controlled Trial of Ceftriaxone and Doxycycline, With or Without Metronidazole, for the Treatment of Acute Pelvic Inflammatory Disease. Clin Infect Dis. 2021 Apr 8;72(7):1181-1189. doi: 10.1093/cid/ciaa101. PMID 32052831

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftriaxone, Doxycycline, Placebo: ceftrixone 250mg IM single dose plus doxycycline 100 mg PO bid x 14 days plus placebo PO bid x 14 days
  ceftriaxone, doxycycline, placebo: ceftrixone 250mg IM single dose plus doxycycline 100 mg PO bid x 14 days plus placebo PO bid x 14 days
- Ceftriaxone, Doxycycline, Metronidazole: ceftriaxone 250 mg IM single dose plus doxycycline 100 mg PO bid x 14 days plus metronidazole 500 mg PO bid x 14 days
  ceftriaxone, doxycycline, metronidazole: ceftriaxone 250 mg IM single dose plus doxycycline 100 mg PO bid x 14 days plus metronidazole 500 mg PO bid x 14 days
Period: Overall Study
Arm/Group | Ceftriaxone, Doxycycline, Placebo | Ceftriaxone, Doxycycline, Metronidazole
Started | 117 | 116
Completed | 113 | 110
Not Completed | 4 | 6
Not completed — Physician Decision | 3 | 3
Not completed — Incarceration | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftriaxone, Doxycycline, Placebo | Ceftriaxone, Doxycycline, Metronidazole | Total
Number analyzed (Participants) | 117 | 116 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (4.3) | 24.7 (5.1) | 24.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 116 | 233
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 106 | 105 | 211
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 76 | 68 | 144
  White | 28 | 35 | 63
  More than one race | 10 | 9 | 19
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 117 | 116 | 233

OUTCOME MEASURES:

1. Primary Outcome: Clearance of Anaerobic Organisms From the Endometrium
Description: Clearance of anaerobic microorganisms from the endometrium at the 30 day follow-up visit among women who had anaerobic microorganisms detected in their endometrial tissue sample at enrollment. Clearance is defined as no anaerobic microorganisms detected in the endometrial tissue biopsy sample collected at the 30-day visit.
Time Frame: Enrollment to 30 days
Population: Women who had anaerobic microorganisms detected in their endometrial biopsy sample at enrollment based on standard bacterial culture techniques.
Measure: Number; unit: participants
Arm/Group | Ceftriaxone, Doxycycline, Placebo | Ceftriaxone, Doxycycline, Metronidazole
Number analyzed (Participants) | 21 | 19
participants
  Clearance of anaerobes | 14 | 18
  Anaerobes detected | 7 | 1
Statistical Analysis 1: Comparison: Ceftriaxone, Doxycycline, Placebo vs Ceftriaxone, Doxycycline, Metronidazole; Test type: Superiority or Other; p = 0.046, Fisher Exact — P-value for proportion of women who had clearance of anaerobic organisms from the endometrium at the 30-day visit

2. Secondary Outcome: The Prevalence of M. Genitalium in the Cervix and Endometrium From Women With Acute PID.
Description: The number of women who had M. genitalium detected in cervical and endometrial biopsy cultures by nucleic acid amplification tests at enrollment.
Time Frame: enrollment
Measure: Number; unit: participants
Arm/Group | Ceftriaxone, Doxycycline, Placebo | Ceftriaxone, Doxycycline, Metronidazole
Number analyzed (Participants) | 117 | 116
participants
  Detected in cervix only | 16 | 12
  Detected in cervix and endometrium | 8 | 5
  Detected in endometrium only | 3 | 2
  Not detected in cervix and endometrium | 90 | 97

3. Secondary Outcome: The Eradication of M. Genitalium From the Lower and Upper Genital Tract Following Antibiotic Therapy for Acute PID.
Description: M. genitalium not detected in the cervical and endometrial cultures by nucleic acid amplification testing at the 30 day visit among women who had M. genitalium detected at either anatomical site at the enrollment visit.
Time Frame: Enrollment to 30 days
Population: There were 34 women who had M. genitalium detected in the cervix or endometrium at enrollment who had test results from the 30-day visit.
Measure: Number; unit: participants
Arm/Group | Ceftriaxone, Doxycycline, Placebo | Ceftriaxone, Doxycycline, Metronidazole
Number analyzed (Participants) | 21 | 13
participants
  Not detected in cervix & endometrium | 8 | 9
  Detected in cervix or endometrium | 13 | 4
Statistical Analysis 1: Comparison: Ceftriaxone, Doxycycline, Placebo vs Ceftriaxone, Doxycycline, Metronidazole; Test type: Superiority or Other; p = 0.16, Fisher Exact — P-value for proportion of women who did not have M. genitalium detected in the cervix or endometrium at the 30-day visit

4. Secondary Outcome: Resolution of Clinical Signs and Symptoms of Acute PID - Intention to Treat Analysis
Description: Clinical response to treatment is improvement (reduction) of the McCormack Scale total score from baseline to day 3 follow-up visit. Participants without a 3-day measure were considered treatment failures.
Time Frame: Enrollment to 3 day follow up visit
Measure: Number; unit: participants
Arm/Group | Ceftriaxone, Doxycycline, Placebo | Ceftriaxone, Doxycycline, Metronidazole
Number analyzed (Participants) | 117 | 116
participants
  Clinical response | 94 | 96
  No response | 23 | 20
Statistical Analysis 1: Comparison: Ceftriaxone, Doxycycline, Placebo vs Ceftriaxone, Doxycycline, Metronidazole; Test type: Superiority or Other; p = 0.74, Fisher Exact — P-value for proportion of women who experienced resolution of clinical signs and symptoms of PID at the 3-day visit

5. Secondary Outcome: Identification of Endometrial Microorganisms Present Obtained From Women With or Without Evidence of Endometritis.
Description: Identification of endometrial microorganisms present obtained from women with or without evidence of endometritis using a combination of culture methods, rRna sequencing and whole genomic sequencing. The aim is to identify the etiology of endometritis.
Time Frame: enrollment
Population: Women who had an endometrial sample that was sufficient for histologic assessment for endometritis.
Measure: Number; unit: participants
Groups:
- Histological Endometritis Present: Women who had endometritis confirmed by histologic assessment for endometritis. Endometritis was defined as >1 plasma cell per 100X microscopic field, was assessed independently by 2 pathologists blinded to the design
- Histological Endometritis Absent: Women who did not have endometritis confirmed by histologic assessment for endometritis
Arm/Group | Histological Endometritis Present | Histological Endometritis Absent
Number analyzed (Participants) | 70 | 138
participants
  Chlamydia trachomatis | 17 | 5
  Neisseria gonorrhoeae | 8 | 2
  Mycoplasma genitalium | 12 | 5
  Haemophilus influenzae | 5 | 1
  Gardnerella vaginalis | 22 | 25
  Atopobium vaginae | 7 | 13
  Anaerobic gram negative rods | 8 | 8
  Anaerobic gram positive cocci | 10 | 11
  Anaerobic gram positive rods | 4 | 11

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Ceftriaxone, Doxycycline, Placebo | Ceftriaxone, Doxycycline, Metronidazole
Serious Adverse Events (participants affected / at risk) | 5/117 | 7/116
Other Adverse Events (participants affected / at risk) | 94/117 | 104/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftriaxone, Doxycycline, Placebo (N=117) | Ceftriaxone, Doxycycline, Metronidazole (N=116)
Ruptured ovarian cyst, pelvic inflammatory disease increased pain (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Paratubal cyst, right (Reproductive system and breast disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Failed outpatient pelvic inflammatory disease treatment (Reproductive system and breast disorders) | 0 | 2
Pelvic pain, increased (Reproductive system and breast disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pelvic floor muscle spasm (Reproductive system and breast disorders) | 0 | 1
Acute pelvic inflammatory disease (Reproductive system and breast disorders) | 0 | 1
Pelvic inflammatory disease, nausea, and vomiting (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftriaxone, Doxycycline, Placebo (N=117) | Ceftriaxone, Doxycycline, Metronidazole (N=116)
Nausea (Gastrointestinal disorders) | 55 (59) | 58 (58)
Vomiting (Gastrointestinal disorders) | 37 (39) | 40 (42)
Diarrhea (Gastrointestinal disorders) | 30 (30) | 39 (40)
Vaginal discharge, abnormal (Reproductive system and breast disorders) | 4 (4) | 9 (9)
Altered taste (Gastrointestinal disorders) | 5 (5) | 8 (8)
Bacterial vaginosis (Infections and infestations) | 8 (8) | 4 (4)
Headache (General disorders) | 10 (10) | 12 (12)
Loose stool (Gastrointestinal disorders) | 9 (9) | 6 (6)
Vaginal itching (Reproductive system and breast disorders) | 7 (7) | 11 (11)
Vulvovaginal candidiasis (Infections and infestations) | 7 (8) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No